CLINICAL TRIAL: NCT04038567
Title: Optimizing a Self-directed Mobile Mindfulness Intervention for Improving Cardiorespiratory Failure Survivors' Psychological Distress
Brief Title: Optimizing a Mobile Mindfulness Intervention for ICU Survivors
Acronym: LIFT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Washington (Other); University of Colorado, Denver (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00100252; 1U01AT009974 (NIH)
Record Dates: First submitted 2019-07-24; First posted 2019-07-31 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Cardiorespiratory Failure
Keywords: cardiorespiratory failure; critical illness; psychological distress; depression; anxiety; post-traumatic stress disorder; intensive care units; adults; mechanical ventilation
MeSH Terms: conditions — Critical Illness; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Factorial experimental trial as part of a multi-phase optimization strategy (MOST) design
Who Masked: Investigator, Outcomes Assessor
Masking Description: PIs and analysts blinded to allocation. Outcomes completed by participants using web-based interface and thus outcomes assessors as such are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- App introduction to intervention (Other): Introduction to intervention via the mobile app itself.
  Interventions: Behavioral: Mobile mindfulness-based training
- Therapist introduction to intervention (Other): Introduction to intervention via a call from the study therapist.
  Interventions: Behavioral: Mobile mindfulness-based training
- Standard dose (Other): Standard dose of meditation time (once a day).
  Interventions: Behavioral: Mobile mindfulness-based training
- High dose (Other): High dose of meditation time (twice a day).
  Interventions: Behavioral: Mobile mindfulness-based training
- App response to symptoms (Other): Mobile app response to elevated psychological distress symptoms during intervention period.
  Interventions: Behavioral: Mobile mindfulness-based training
- Therapist response to symptoms (Other): Therapist call in response to elevated psychological distress symptoms during intervention period.
  Interventions: Behavioral: Mobile mindfulness-based training

INTERVENTIONS:
Behavioral: Mobile mindfulness-based training — The intervention core is a mobile app-based mindfulness training program designed to be used over a 1-month period. All 6 factorial groups will use the app, though the delivery of the app and response to psychological distress symptoms over time will differ by group.

SUMMARY:
This is a factorial experimental trial involving adult survivors of cardiorespiratory failure treated in intensive care units (ICUs) that is conceptualized as the Optimization Phase of a multiphase optimization strategy (MOST) framework. This will allow optimization of a mobile mindfulness intervention by comparing eight different iterations across domains including impact on symptoms, feasibility, acceptability, usability, scalability, and cost.

DETAILED DESCRIPTION:
As survival has improved for the 2 million people with cardiorespiratory failure managed annually in US intensive care units (ICUs), it has become apparent that these patients suffer from severe and persistent post-discharge symptoms of psychological distress including depression, anxiety, and post-traumatic stress disorder (PTSD). However, few targeted interventions exist that are relevant to patients' experiences and that accommodate their many physical, social, and financial barriers to personalized care. To fill this gap, an innovative app-based mobile mindfulness training program twas developed hat promotes automated care delivery and self-management of symptom-related distress.

Subsequently, a pilot randomized clinical trial (RCT) called the LIFT study (R34 AT00819) compared mobile mindfulness to both a standard telephone mindfulness program and an ICU education control among survivors of cardiorespiratory failure. Key findings were that mobile mindfulness was feasibly delivered, acceptable, usable, and had a greater clinical impact on psychological distress than either comparator. This trial also highlighted opportunities to improve the intervention's impact related to its targeted population, content delivery, and system technology.

To address these gaps, this 5-year project is conceptualized as the Optimization Phase of a multiphase optimization strategy (MOST) framework. It will optimize mobile mindfulness with four specific aims as described in the following sections. At the conclusion of this factorial randomized clinical trial study involving 240 cardiorespiratory failure survivors, a mobile mindfulness system fully optimized for usability, efficiency, scalability, and clinical impact will be delivered that will be off-the-shelf ready for a next-step definitive RCT-and can serve as a model for distance-based mind and body interventions.

ELIGIBILITY:
INCLUSION CRITERIA

1. Adult (age ≥18)
2. Acute cardiorespiratory failure:

   * Acute respiratory failure, defined as ≥1 of the following:
   * mechanical ventilation via endotracheal tube for ≥12 hours
   * non-invasive ventilation (CPAP, BiPAP) for ≥4 hours in a 24-hour period provided for acute respiratory failure in an ICU (not for obstructive sleep apnea or other stable use)
   * high flow nasal cannula or face mask oxygen for ≥4 hours in a 24-hour period and / or
   * Acute cardiac / circulatory failure, defined as ≥1 of the following:
   * use of vasopressors for shock of any etiology for ≥1 hour
   * use of inotropes for shock of any etiology for ≥1 hour
   * use of pulmonary vascular vasoactive medications
   * use of aortic balloon pump for cardiogenic shock for ≥1 hour
3. Managed in an adult medical cardiac, trauma, surgical, or neurological ICU, stepdown unit, or monitored ward unit for ≥24 hours during the time inclusion criterion #2 is met.
4. Cognitive status intact

   * No history of pre-existing significant cognitive impairment (e.g., dementia) as per medical chart
   * Absence of current significant cognitive impairment (impairment defined as ≥3 errors on the Callahan cognitive status screen)
   * Decisional capacity present
5. Absence of severe and/or persistent mental illness

   * Treatment for severe and/or persistent mental illness (e.g., psychosis, bipolar affective disorder, schizoaffective disorder, schizoid personality disorder, schizophrenia [as per medical record], hospitalization for any psychiatric disorder) within the 6 months preceding the current hospital admission
   * No endorsement of suicidality at time of admission or informed consent
   * No active substance abuse within the 3 months preceding the current admission serious enough to limit completion of study procedures in the opinion of the site investigator.
6. English fluency.

EXCLUSION CRITERIA (in hospital):

1. Hospitalized within the preceding 3 months with life-threatening illness or injury.

   Patients may be enrolled into the study if they had a hospitalization within the preceding 3 months that is determined to be non-serious. Non-serious admissions are defined as those admissions that are non-life threatening and/or potentially impacting patient's well-being long-term or likely to precipitate additional future admissions. Examples of non-life-threatening hospitalizations could be, but may not be limited to, admission for a bronchoscopy, admission for deep vein thrombosis, or admission to ED resulting in overnight stay for cardiac work-up.
2. Admitted from a location other than home (e.g., nursing home, long-term acute care facility, inpatient rehabilitation facility)
3. Anticipated or actual discharge to a location other than independent in a home setting (e.g., nursing home, long-term acute care facility, inpatient rehabilitation facility, home hospice)
4. Complex medical care expected soon after discharge (e.g., planned surgeries, transplantation evaluation, extensive travel needs for hemodialysis, disruptive chemotherapy/radiation regimen)
5. Unable to complete study procedures as determined by staff
6. Lack of reliable smartphone with cellular data plan or wifi access

   EXCLUSION CRITERIA (at T1, post-discharge):
7. Low baseline psychological distress symptoms, defined as the absence of the following at T1: PHQ-9 score <5
8. Failure to randomize within 2 month (60 days) post-discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Cox, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - University of Colorado - Denver, Aurora, Colorado
  - Duke University Medical Center, Durham, North Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will follow NIH/NCCIH guidelines for data access.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We will follow NIH and institutional guidelines.
Access Criteria: We will follow NIH and institutional guidelines. Given the length of time that will elapse during the study, we will need to adhere to the rules present at that time.

REFERENCES:
- [Background] Cox CE, Porter LS, Buck PJ, Hoffa M, Jones D, Walton B, Hough CL, Greeson JM. Development and preliminary evaluation of a telephone-based mindfulness training intervention for survivors of critical illness. Ann Am Thorac Soc. 2014 Feb;11(2):173-81. doi: 10.1513/AnnalsATS.201308-283OC. PMID 24303911
- [Background] Cox CE, Hough CL, Jones DM, Ungar A, Reagan W, Key MD, Gremore T, Olsen MK, Sanders L, Greeson JM, Porter LS. Effects of mindfulness training programmes delivered by a self-directed mobile app and by telephone compared with an education programme for survivors of critical illness: a pilot randomised clinical trial. Thorax. 2019 Jan;74(1):33-42. doi: 10.1136/thoraxjnl-2017-211264. Epub 2018 May 23. PMID 29793970
- [Background] Cox CE, Olsen MK, Gallis JA, Porter LS, Greeson JM, Gremore T, Frear A, Ungar A, McKeehan J, McDowell B, McDaniel H, Moss M, Hough CL. Optimizing a self-directed mobile mindfulness intervention for improving cardiorespiratory failure survivors' psychological distress (LIFT2): Design and rationale of a randomized factorial experimental clinical trial. Contemp Clin Trials. 2020 Sep;96:106119. doi: 10.1016/j.cct.2020.106119. Epub 2020 Aug 15. PMID 32805434
- [Derived] Cox CE, Gallis JA, Olsen MK, Porter LS, Gremore T, Greeson JM, Morris C, Moss M, Hough CL. Mobile Mindfulness Intervention for Psychological Distress Among Intensive Care Unit Survivors: A Randomized Clinical Trial. JAMA Intern Med. 2024 Jul 1;184(7):749-759. doi: 10.1001/jamainternmed.2024.0823. PMID 38805199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note that this is a factorial experimental trial in which 3 factors were examined, each at 2 levels (i.e., a 2^3 design).
  In this trial the 3 factors and 2 levels are as follows:
  1. Introduction to intervention (app introduction vs. therapist introduction)
  2. Dose (standard vs. high)
  3. Response to depression symptoms that increase during the intervention period (app response vs. therapist response)
Groups:
- App Introduction to Intervention, High Dose, and Therapist Response: Introduction to intervention via the mobile app itself. High dose of meditation time (twice a day). Therapist call in response to elevated psychological distress symptoms during intervention period.
- Therapist Introduction to Intervention, High Dose, and Therapist Response: Introduction to intervention via a call from the study therapist. High dose of meditation time (twice a day). Therapist call in response to elevated psychological distress symptoms during intervention period.
- App Introduction to Intervention, Standard Dose, and Therapist Response: Introduction to intervention via the mobile app itself. Standard dose of meditation time (once a day). Therapist call in response to elevated psychological distress symptoms during intervention period.
- Therapist Introduction to Intervention, Standard Dose, and Therapist Response: Introduction to intervention via a call from the study therapist. Standard dose of meditation time (once a day). Therapist call in response to elevated psychological distress symptoms during intervention period.
- App Introduction to Intervention, High Dose, and App Response: Introduction to intervention via the mobile app itself. High dose of meditation time (twice a day). Mobile app response to elevated psychological distress symptoms during intervention period.
- Therapist Introduction to Intervention, High Dose, and App Response: Introduction to intervention via a call from the study therapist. High dose of meditation time (twice a day). Mobile app response to elevated psychological distress symptoms during intervention period.
- App Introduction to Intervention, Standard Dose, and App Response: Introduction to intervention via the mobile app itself. Standard dose of meditation time (once a day). Mobile app response to elevated psychological distress symptoms during intervention period.
- Therapist Introduction to Intervention, Standard Dose, and App Response: Introduction to intervention via a call from the study therapist. Standard dose of meditation time (once a day). Mobile app response to elevated psychological distress symptoms during intervention period.
Period: Overall Study
Arm/Group | App Introduction to Intervention, High Dose, and Therapist Response | Therapist Introduction to Intervention, High Dose, and Therapist Response | App Introduction to Intervention, Standard Dose, and Therapist Response | Therapist Introduction to Intervention, Standard Dose, and Therapist Response | App Introduction to Intervention, High Dose, and App Response | Therapist Introduction to Intervention, High Dose, and App Response | App Introduction to Intervention, Standard Dose, and App Response | Therapist Introduction to Intervention, Standard Dose, and App Response
Started | 30 | 31 | 31 | 32 | 32 | 31 | 30 | 30
Completed | 21 | 23 | 23 | 25 | 19 | 24 | 22 | 25
Not Completed | 9 | 8 | 8 | 7 | 13 | 7 | 8 | 5
Not completed — Lost to Follow-up | 6 | 4 | 5 | 4 | 6 | 4 | 4 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1 | 4 | 1 | 1 | 1
Not completed — missed survey window | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 2
Not completed — technical issues | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Medical issues (i.e., illness) | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | App Introduction to Intervention, High Dose, and Therapist Response | Therapist Introduction to Intervention, High Dose, and Therapist Response | App Introduction to Intervention, Standard Dose, and Therapist Response | Therapist Introduction to Intervention, Standard Dose, and Therapist Response | App Introduction to Intervention, High Dose, and App Response | Therapist Introduction to Intervention, High Dose, and App Response | App Introduction to Intervention, Standard Dose, and App Response | Therapist Introduction to Intervention, Standard Dose, and App Response | Total
Number analyzed (Participants) | 30 | 31 | 31 | 32 | 32 | 31 | 30 | 30 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (15.0) | 51.6 (14.6) | 48.2 (15.7) | 48.8 (14.8) | 47.4 (16.4) | 49.4 (17.1) | 51.3 (14.4) | 49.4 (15.2) | 50.22 (15.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 13 | 15 | 10 | 16 | 16 | 11 | 104
  Male | 18 | 20 | 18 | 17 | 22 | 15 | 14 | 19 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 3 | 1 | 4 | 5 | 4 | 24
  Not Hispanic or Latino | 26 | 29 | 29 | 27 | 30 | 26 | 24 | 26 | 217
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 5
  Asian | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Black or African American | 5 | 4 | 4 | 3 | 8 | 6 | 4 | 1 | 35
  White | 21 | 24 | 24 | 25 | 17 | 24 | 21 | 23 | 179
  More than one race | 3 | 0 | 2 | 2 | 1 | 0 | 3 | 1 | 12
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 4 | 1 | 2 | 1 | 10
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 31 | 32 | 32 | 31 | 30 | 30 | 247

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire-9 Item Scale (PHQ-9)
Description: Absolute values, not change scores. Depression symptoms. Scores range from 0 (better) to 27 (worse)
Time Frame: 1 month post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- App Response: Mobile app response to elevated psychological distress symptoms during intervention period.
- Therapist Response: Therapist call in response to elevated psychological distress symptoms during intervention period.
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 91 | 100 | 97 | 94 | 92 | 99
units on a scale | 6.2 (4.7) | 6.4 (4.8) | 7.0 (5.2) | 5.6 (4.2) | 6.2 (5.3) | 6.4 (4.3)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; Values are change in model-estimated means for therapist vs. app introduction. Intervention components are coded as follows: introduction method (therapist [1] vs app [-1]), dose (high [1] vs low [-1]), and symptom management (therapist [1] vs app [-1]); Test type: Superiority; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-1.14 to 1.20]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; Values are change in model-estimated means for his vs. standard dose. Intervention components are coded as follows: introduction method (therapist [1] vs app [-1]), dose (high [1] vs low [-1]), and symptom management (therapist [1] vs app [-1]); Test type: Superiority; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-2.39 to -0.04]
Statistical Analysis 3: Comparison: App Response vs Therapist Response; Values are change in model-estimated means for therapist vs. app response. Intervention components are coded as follows: introduction method (therapist [1] vs app [-1]), dose (high [1] vs low [-1]), and symptom management (therapist [1] vs app [-1]); Test type: Superiority; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-1.12 to 1.23]

2. Secondary Outcome: Generalized Anxiety Disorder 7-item Scale (GAD-7)
Description: Absolute values, not change scores. Anxiety symptoms. Scores range from 0 (better) to 21 (worse)
Time Frame: Between baseline 1 month post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 87 | 95 | 95 | 87 | 88 | 94
units on a scale | 5.5 (5.4) | 4.9 (4.5) | 6.2 (5.3) | 4.2 (4.3) | 5.1 (4.7) | 5.3 (5.1)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -1.14, 95% CI 2-sided [-2.12 to -0.16]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; Values are change in model-estimated means for high vs. standard dose. Intervention components are coded as follows: introduction method (therapist [1] vs app [-1]), dose (high [1] vs low [-1]), and symptom management (therapist [1] vs app [-1]); Test type: Superiority; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.80 to 1.49]
Statistical Analysis 3: Comparison: App Response vs Therapist Response; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.48 to 1.49]

3. Secondary Outcome: Patient Health Questionnaire-9 Item Scale (PHQ-9)
Description: Absolute values, not change scores. Depression symptoms. Scores range from 0 (better) to 27 (worse)
Time Frame: Between baseline 3 months post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response to Symptoms | Therapist Response to Symptoms
Number analyzed (Participants) | 87 | 95 | 95 | 87 | 88 | 94
units on a scale | 7.28 (5.76) | 7.04 (5.50) | 8.12 (6.23) | 6.10 (4.65) | 6.73 (5.69) | 7.55 (5.53)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-1.66 to 1.01]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = -1.47, 95% CI 2-sided [-2.81 to -0.14]
Statistical Analysis 3: Comparison: App Response to Symptoms vs Therapist Response to Symptoms; Values are change in model-estimated means for therapist vs. app response to symptoms. Intervention components are coded as follows: introduction method (therapist [1] vs app [-1]), dose (high [1] vs low [-1]), and symptom management (therapist [1] vs app [-1]); Test type: Superiority; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-0.52 to 2.15]

4. Secondary Outcome: Generalized Anxiety Disorder 7-item Scale (GAD-7)
Description: Absolute values, not change scores. Anxiety symptoms. Scores range from 0 (better) to 21 (worse)
Time Frame: Between baseline 3 months post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 87 | 95 | 95 | 87 | 88 | 94
units on a scale | 5.62 (5.07) | 5.69 (5.28) | 6.83 (5.74) | 4.38 (4.12) | 6.25 (5.45) | 5.11 (4.86)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; Test type: Superiority; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-1.23 to 0.91]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; Test type: Superiority; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-2.29 to -0.15]
Statistical Analysis 3: Comparison: App Response vs Therapist Response; Test type: Superiority; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.77 to 0.37]

5. Secondary Outcome: Post-Traumatic Stress Symptom Inventory (PTSS)
Description: Absolute values, not change scores. PTSD symptoms. Scores can range from 10 (best) to 70 (worst).
Time Frame: Between baseline 3 months post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 87 | 95 | 95 | 87 | 88 | 94
units on a scale | 29.94 (23.88) | 27.83 (15.10) | 31.75 (24.05) | 25.67 (13.05) | 29.75 (23.95) | 27.99 (14.89)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-4.41 to 1.25]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; Values are change in model-estimated means for hig vs. standard dose. Intervention components are coded as follows: introduction method (therapist [1] vs app [-1]), dose (high [1] vs low [-1]), and symptom management (therapist [1] vs app [-1]); Test type: Superiority; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-3.26 to 2.42]
Statistical Analysis 3: Comparison: App Response vs Therapist Response; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Mean Difference (Final Values) = 1.49, 95% CI 2-sided [-1.35 to 4.33]

6. Secondary Outcome: Intervention Adherence: Activity in App During Final Week of Intervention
Description: Quantified by number with activity (or not) in app during final week (4) of intervention
Time Frame: 1 month post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 125 | 122 | 124 | 120 | 123 | 124
Participants | 105 | 108 | 112 | 104 | 105 | 111

7. Secondary Outcome: Intervention Adherence: Number of Views of Content
Description: Quantified by mean (SD) number of intervention content (audio, video, text) views
Time Frame: 1 month post-randomization
Measure: Mean (Standard Deviation); unit: mobile app content views
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 125 | 122 | 124 | 120 | 123 | 124
mobile app content views | 34.24 (31.37) | 40.03 (35.82) | 34.88 (35.81) | 39.38 (31.38) | 40.53 (38.31) | 33.70 (28.14)

8. Secondary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: A measure of acceptability. Scores can range from 8 (worst) to 32 (best)
Time Frame: 3 months post-randomization
Population: Data not collected.
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response to Symptoms | Therapist Response to Symptoms
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Systems Usability Scale (SUS)
Description: A measure of intervention usability. Each of 10 items is scored from 1 to 5. For each of the odd numbered questions, subtract 1 from the score.
  For each of the even numbered questions, subtract their value from 5. Take these new values and add up the total score. Then multiply this by 2.5.Scores can range from 0 (worst) to 100 (best)
Time Frame: 3 months post-randomization
Population: Data not collected.
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response to Symptoms | Therapist Response to Symptoms
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Mindful Attention Awareness Scale (MAAS)
Description: This is the absolute value, not change score. A measure of mindfulness qualities. Scores can range from 5 (worst) to 30 (best).
Time Frame: Between baseline and 1 month post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 91 | 100 | 97 | 94 | 92 | 99
units on a scale | 23.41 (5.22) | 23.49 (5.61) | 22.86 (5.06) | 24.04 (5.71) | 23.31 (5.67) | 23.59 (5.18)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-0.62 to 1.78]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = 0.73, 95% CI 2-sided [-0.47 to 1.92]
Statistical Analysis 3: Comparison: App Response vs Therapist Response; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-1.00 to 1.39]

11. Secondary Outcome: Mindful Attention Awareness Scale (MAAS)
Description: These are absolute values, not change scores. A measure of mindfulness qualities. Scores can range from 5 (worst) to 30 (best).
Time Frame: Between baseline 3 months post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 87 | 95 | 95 | 87 | 88 | 94
units on a scale | 22.43 (5.51) | 23.03 (6.17) | 22.43 (5.79) | 23.08 (5.94) | 22.57 (6.23) | 22.90 (5.51)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [-0.45 to 2.27]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-1.33 to 1.38]
Statistical Analysis 3: Comparison: App Response vs Therapist Response; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.72 to 0.99]

12. Secondary Outcome: Patient Health Questionnaire 10-item Scale (PHQ-10)
Description: These are absolute values, not change scores. An adapted version of the PHQ-15; a measure of physical symptoms. Scores can range from 10 (best) to 20 (worst).
Time Frame: Between baseline and 1 month post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 91 | 100 | 97 | 94 | 92 | 99
units on a scale | 6.50 (3.16) | 6.19 (3.45) | 6.66 (3.44) | 6.02 (3.16) | 6.31 (3.32) | 6.37 (3.32)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.30 to 0.30]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.33 to 0.27]
Statistical Analysis 3: Comparison: Standard Dose vs High Dose; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-.55 to 1.05]

13. Secondary Outcome: Patient Health Questionnaire 10-item Scale (PHQ-10)
Description: This is an absolute value, not a change score. An adapted version of the PHQ-15; a measure of physical symptoms. Scores can range from 10 (best) to 20 (worst).
Time Frame: Between baseline 3 months post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 95 | 87 | 87 | 95 | 88 | 94
units on a scale | 6.21 (3.44) | 5.63 (3.72) | 6.15 (3.86) | 5.64 (3.28) | 5.85 (3.58) | 5.96 (3.62)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; Test type: Superiority; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.41 to 0.41]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; Test type: Superiority; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.27 to 0.55]
Statistical Analysis 3: Comparison: App Response vs Therapist Response; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.40 to 1.42]

14. Secondary Outcome: EuroQOL Scale
Description: This is an absolute, not change, value. the EuroQOL is a measure of quality of life. Scores can range from 0 (worst) to 100 (best)
Time Frame: Between baseline and 1 month post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 91 | 100 | 97 | 94 | 92 | 99
units on a scale | 61.56 (23.07) | 63.60 (21.25) | 58.87 (21.98) | 66.56 (21.64) | 63.91 (21.43) | 61.43 (22.75)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 2.33, 95% CI 2-sided [-3.25 to 7.91]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = 4.82, 95% CI 2-sided [-0.76 to 10.40]
Statistical Analysis 3: Comparison: App Response vs Therapist Response; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-5.60 to 5.56]

15. Secondary Outcome: Change in EuroQOL Scale
Description: A measure of quality of life. Scores can range from 0 (worst) to 100 (best)
Time Frame: Between baseline 3 months post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 91 | 100 | 97 | 94 | 92 | 99
units on a scale | 62.07 (22.23) | 65.47 (24.44) | 61.68 (24.15) | 66.21 (22.48) | 65.02 (24.87) | 62.74 (22.03)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 3.18, 95% CI 2-sided [-3.01 to 9.37]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = 1.28, 95% CI 2-sided [-4.92 to 7.47]
Statistical Analysis 3: Comparison: App Response vs Therapist Response; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-6.09 to 6.30]

16. Secondary Outcome: Distress Associated With Depression Symptom Frequency
Description: A visual analog scale appended to the PHQ-9 which allows participants to report how distressing they perceive the depression symptoms to be that they reported in the PHQ-9. Scores range from 0 (best) to 100 (worst)
Time Frame: Between baseline and 1 month post-randomization; THIS WAS NOT RECORDED
Population: Data were not collected
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Distress Associated With Depression Symptom Frequency
Description: as for outcome 16
Time Frame: At 1 month post-randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 91 | 100 | 97 | 94 | 92 | 99
units on a scale | 41.22 (28.53) | 37.40 (26.65) | 44.26 (28.96) | 34.02 (25.14) | 41.34 (28.36) | 37.25 (26.78)

18. Secondary Outcome: Distress Associated With Anxiety Symptom Frequency
Description: A visual analog scale appended to the GAD-7 which allows participants to report how distressing they perceive the depression symptoms to be that they reported in the GAD-7. Scores range from 0 (best) to 100 (worst)
Time Frame: At 1 month post-randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 125 | 122 | 124 | 123 | 123 | 124
units on a scale | 45.31 (26.50) | 49.54 (25.04) | 50.11 (26.07) | 44.67 (25.38) | 48.57 (24.47) | 46.24 (27.15)

19. Secondary Outcome: Distress Associated With Anxiety Symptom Frequency
Description: as for outcome 18
Time Frame: Between baseline 3 months post-randomization
Population: Data were not collected
Arm/Group | High Dose
Number analyzed (Participants) | 0

20. Secondary Outcome: Distress Associated With PTSD Symptom Frequency
Description: A visual analog scale appended to the PTSS which allows participants to report how distressing they perceive the depression symptoms to be that they reported in the PTSS. Scores range from 0 (best) to 100 (worst)
Time Frame: At 1 month post-randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 125 | 122 | 124 | 123 | 123 | 124
units on a scale | 44.60 (30.52) | 47.04 (29.04) | 49.56 (28.59) | 42.02 (30.54) | 47.69 (28.63) | 43.94 (30.84)

21. Secondary Outcome: Distress Associated With PTSD Symptom Frequency
Description: Absolute values, not change scores. A visual analog scale appended to the PTSS which allows participants to report how distressing they perceive the depression symptoms to be that they reported in the PTSS. Scores range from 0 (best) to 100 (worst)
Time Frame: At 3 months post-randomization
Population: Data were not collected
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Post-Traumatic Stress Symptom Inventory (PTSS)
Description: Absolute values, not change scores. Post-traumatic stress disorder symptoms. Scores can range from 10 (best) to 70 (worst).
Time Frame: Between baseline and 1 month post-randomization
Population: Participants who had data collected at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 91 | 100 | 97 | 94 | 92 | 99
units on a scale | 28.91 (28.14) | 26.38 (13.08) | 31.53 (28.04) | 23.65 (11.04) | 29.53 (27.81) | 25.77 (13.36)
Statistical Analysis 1: Comparison: App Introduction to Intervention vs Therapist Introduction to Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -2.70, 95% CI 2-sided [-5.26 to -0.13]
Statistical Analysis 2: Comparison: Standard Dose vs High Dose; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = -1.89, 95% CI 2-sided [-4.46 to 0.67]
Statistical Analysis 3: Comparison: App Response vs Therapist Response; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-3.31 to 1.83]

23. Secondary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: A measure of acceptability. Scores can range from 8 (worst) to 32 (best)
Time Frame: 1 month post-randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response | Therapist Response
Number analyzed (Participants) | 91 | 100 | 97 | 94 | 92 | 99
units on a scale | 25.27 (4.46) | 25.31 (4.82) | 24.86 (5.11) | 25.71 (4.10) | 25.81 (4.58) | 24.79 (4.67)

24. Secondary Outcome: Systems Usability Scale (SUS)
Description: as for outcome 9
Time Frame: 1 month post-randomization
Population: Data not collected.
Arm/Group | App Introduction to Intervention | Therapist Introduction to Intervention | Standard Dose | High Dose | App Response to Symptoms | Therapist Response to Symptoms
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events:
  1. death
  2. hospitalization for any reason
  3. Suicidal ideation as indicated by a response on the PHQ-9 item 9 as any response other than 0 ('never')
Arm/Group | App Introduction to Intervention, High Dose, and Therapist Response | Therapist Introduction to Intervention, High Dose, and Therapist Response | App Introduction to Intervention, Standard Dose, and Therapist Response | Therapist Introduction to Intervention, Standard Dose, and Therapist Response | App Introduction to Intervention, High Dose, and App Response | Therapist Introduction to Intervention, High Dose, and App Response | App Introduction to Intervention, Standard Dose, and App Response | Therapist Introduction to Intervention, Standard Dose, and App Response
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31 | 0/31 | 1/32 | 1/32 | 0/31 | 0/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 6/30 | 4/31 | 1/31 | 2/32 | 3/32 | 5/31 | 2/30 | 2/30
Other Adverse Events (participants affected / at risk) | 0/30 | 1/31 | 1/31 | 1/32 | 1/32 | 1/31 | 1/30 | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | App Introduction to Intervention, High Dose, and Therapist Response (N=30) | Therapist Introduction to Intervention, High Dose, and Therapist Response (N=31) | App Introduction to Intervention, Standard Dose, and Therapist Response (N=31) | Therapist Introduction to Intervention, Standard Dose, and Therapist Response (N=32) | App Introduction to Intervention, High Dose, and App Response (N=32) | Therapist Introduction to Intervention, High Dose, and App Response (N=31) | App Introduction to Intervention, Standard Dose, and App Response (N=30) | Therapist Introduction to Intervention, Standard Dose, and App Response (N=30)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 1 (8) | 2 (2) | 3 (3) | 5 (5) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | App Introduction to Intervention, High Dose, and Therapist Response (N=30) | Therapist Introduction to Intervention, High Dose, and Therapist Response (N=31) | App Introduction to Intervention, Standard Dose, and Therapist Response (N=31) | Therapist Introduction to Intervention, Standard Dose, and Therapist Response (N=32) | App Introduction to Intervention, High Dose, and App Response (N=32) | Therapist Introduction to Intervention, High Dose, and App Response (N=31) | App Introduction to Intervention, Standard Dose, and App Response (N=30) | Therapist Introduction to Intervention, Standard Dose, and App Response (N=30)
Suicidal ideation (per PHQ-9 item 9) (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) — Anyone responding to PHQ-9 item 9 with a response other than '0' to question regarding suicidal ideation. This survey was done 5-6 times on every participant during the trial, so it is a sum of all these events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT04038567/Prot_001.pdf
  • Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT04038567/SAP_002.pdf
  • Informed Consent Form (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT04038567/ICF_000.pdf